CLINICAL TRIAL: NCT02453750
Title: Investigation of Airway Inflammation in Congenital Diaphragmatic Hernia Patients
Brief Title: Airway Inflammation in Congenital Diaphragmatic Hernia Patients
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: The Hospital for Sick Children (Other)
Responsible Party: Principal Investigator, Theo Moraes, Staff Respirologist, The Hospital for Sick Children
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 1000028032
Record Dates: First submitted 2015-05-21; First posted 2015-05-25 (Estimated); Results first posted 2019-01-31 (Actual); Last update posted 2019-01-31 (Actual); Status verified 2018-08

CONDITIONS: Congenital Diaphragmatic Hernia
Keywords: Congenital Diaphragmatic Hernia; Airway Inflammation; Asthma; Hypersaline; Pediatrics
MeSH Terms: conditions — Hernias, Diaphragmatic, Congenital; Asthma

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Hypersaline and Bronchodilator Response (Experimental): After the subject has performed post-bronchodilator spirometry, they will inhale 5 mls of 3% hypertonic saline for 7 minutes by nebulizer.
  Interventions: Drug: Hypersaline; Drug: Bronchodilator Response

INTERVENTIONS:
Drug: Hypersaline — Subject will inhale 5 mls of 3% hypertonic saline for 7 minutes by nebulizer. Sputum production (with cough) will be attempted post inhalation. A maximum of 3 hypertonic saline inhalations will be attempted if inhalation does not generate a productive cough. If sputum induction is not successful and the FEV1 falls <10%, the concentration of inhaled hypertonic saline will increase from 3 to 4%. If 5 mls of 4% hypertonic saline inhaled for 7 minutes does not produce a productive cough we will proceed to 5%. If 5 mls of 5% hypertonic saline inhaled for 7 minutes does not produce a productive cough the test is complete and the sample is labelled 'no sputum collected'. If FEV1 falls >10%, the previous step will be repeated.
Drug: Bronchodilator Response — A bronchodilator (Salbutamol 200 mcg or 2 puffs inhaled via spacer device) will be administered to all subjects in the pulmonary function laboratory. 15 minutes after administration of the bronchodilator spirometry will be repeated. This is performed routinely in CDH clinic and is not an additional test for this study.

SUMMARY:
We propose to examine Congenital Diaphragmatic Hernia (CDH) patients for evidence of airway inflammation as a first step to characterize the reported bronchodilator responsiveness. Airway biopsy studies are invasive and thus we propose to perform induced sputum studies to document the amount and type of inflammation present. Another ancillary non-invasive measure of airway inflammation that we will use is exhaled nitric oxide (NO). The primary objective of this study is to determine if CDH patients have any evidence of airway inflammation. The hypothesis of this study is that children with CDH do not have evidence of airway inflammation associated with bronchodilator responsiveness. Based on this information, treatment for CDH patients will hopefully be more accurate and appropriate for their specific needs.

ELIGIBILITY:
Inclusion Criteria:

* 6 - 18 years of age at enrolment
* Clinically stable at enrolment
* Attending follow-up in the CDH Clinic at SickKids

Exclusion Criteria:

* Unable to perform pulmonary function testing
* Clinically unstable at enrolment
* Known hypersensitivity to salbutamol

Ages: 6 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 21 (Actual)
Dates: Start 2012-02; Primary Completion 2013-10 (Actual); Study Completion 2013-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Theo Moraes, MD, Principal Investigator — The Hospital for Sick Children
Locations (1):
- The Hospital for Sick Children, Toronto, Ontario, Canada

RESULTS

PARTICIPANT FLOW:
Groups:
- Hypersaline and Bronchodilator Response: Each child will perform a sputum induction to obtain cells for analysis.
Period: Overall Study
Arm/Group | Hypersaline and Bronchodilator Response
Started | 21
Completed | 21
Not Completed | 0

BASELINE CHARACTERISTICS:
Groups:
- Hypersaline and Bronchodilator Response: After the subject has performed post-bronchodilator spirometry, they will inhale 5 mls of 3% hypertonic saline for 7 minutes by nebulizer to obtain cells for analysis.
Arm/Group | Hypersaline and Bronchodilator Response
Number analyzed (Participants) | 21
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 21
  Between 18 and 65 years | 0
  >=65 years | 0
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 7
  Male | 14
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Elevated Sputum Eosinophils
Description: Number of participants with sputum eosinophils greater than 3% percent of cells in the sputum
Time Frame: post sputum induction
Population: 15 gave reasonable sputum for analysis, none had elevated sputum eosinophils
Measure: Number; unit: participants
Groups:
- Hypersaline and Bronchodilator Response: everyone performs sputum induction
Arm/Group | Hypersaline and Bronchodilator Response
Number analyzed (Participants) | 15
participants | 0

2. Secondary Outcome: Number of Participant With Elevated Sputum Neutrophils
Description: Elevation is defined as sputum neutrophils > or = 61% neutrophils = neutrophilic inflammation
Time Frame: Baseline, +30 minutes
Population: 15 gave reasonable sputum
Measure: Number; unit: participants
Arm/Group | Hypersaline and Bronchodilator Response
Number analyzed (Participants) | 15
participants | 0

3. Secondary Outcome: Number of Participant With Elevated Exhaled Nitric Oxide (NO) Level
Description: exhaled NO measurements will be performed according to the American Thoracic Society and European Respiratory Society guidelines. These tests are performed routinely as part of the respiratory evaluation of these patients and are not additional tests added for this study.
  greater than 20 ppb was considered elevated
Time Frame: 30 min
Population: only 12 performed eNO
Measure: Count of Participants; unit: Participants
Groups:
- Hypersaline and Bronchodilator Response: eNO measured
Arm/Group | Hypersaline and Bronchodilator Response
Number analyzed (Participants) | 12
Participants | 2

4. Secondary Outcome: Number of Participant With Bronchodilator Response
Description: defined as a = or > 12% change in FEV1 post bronchodilator
Time Frame: life time of child (age 6 to present age)
Population: all subjects performed PFTs
Measure: Number; unit: participants
Groups:
- Hypersaline and Bronchodilator Response: spiro performed at start of visit
Arm/Group | Hypersaline and Bronchodilator Response
Number analyzed (Participants) | 21
participants | 15

ADVERSE EVENTS:
Arm/Group | Hypersaline and Bronchodilator Response
All-Cause Mortality (participants affected / at risk) | 0/21
Serious Adverse Events (participants affected / at risk) | 0/21
Other Adverse Events (participants affected / at risk) | 0/21

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No